CLINICAL TRIAL: NCT03604055
Title: Can we Prevent Recurrences in the Endoscopic Treatment of Endobronchial Hamartomas?
Brief Title: Can Recurrence of Hamartomas be Prevented?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Zafer Aktaş, Principal Investigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Za1238
Record Dates: First submitted 2018-07-11; First posted 2018-07-27 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Airway Obstruction; Hamartoma of Lung
Keywords: Hamartoma, Cryotherapy
MeSH Terms: conditions — Airway Obstruction; Hamartoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endobronchial hamartomas treatment (Other): After removal of endobronchial lesions, cryotherapy is applied to the area of origin. Recurrences are followed. Recurrences are recorded as poor results, compared with good results.
  Interventions: Procedure: Endobronchial hamartomas treatment

INTERVENTIONS:
Procedure: Endobronchial hamartomas treatment — General anesthesia was administered by an intravenous anesthesia technique. Patients were intubated with a rigid bronchoscope. Debulking procedures were performed by mechanical tumor resection (MTR) using the tip of the rigid bronchoscope, rigid pliers or argon plasma coagulation assisted MTR or cryorecanalization or electrocautery - snare probe. An innovation of our study was that cryotherapy was performed in the regions where the lesions originated after debulking

SUMMARY:
Background. Recently, treatment of endobronchial hamartomas with interventional bronchoscopic methods has become possible. Although there are several reports of therapeutic benefits, the protocol of administration varies between centers and high recurrence rates continue to be a problem. In this study, the investigators aimed to show that cryotherapy applied to the root of the bronchial wall after removal of the intraluminal portion of endobronchial hamartoma with interventional bronchoscopic methods can prevent recurrences.

Methods. Between 2012 and 2016, the treatment outcomes and long-term follow-up data of 21 consecutive patients with symptomatic endobronchial hamartomas treated by interventional bronchoscopic methods were prospectively recorded. After debulking, cryotherapy was applied to the root of the bronchial wall of all lesions. The data were analyzed retrospectively.

DETAILED DESCRIPTION:
Introduction:

Hamartomas are the most common benign pulmonary tumors. The incidence varies between 0.025% and 0.032%. Endobronchial hamartomas constitute 10-20% of all pulmonary hamartomas. Pulmonary hamartomas are usually asymptomatic and are diagnosed incidentally. In endobronchial hamartomas, at least one of the symptoms of airway obstruction such as cough, hemoptysis and dyspnea are most commonly seen (80%). The results of bronchoscopic removal of symptomatic endobronchial hamartomas and recurrence rates have been the subject of several studies.

Cryotherapy is an endobronchial therapy based on the cytotoxic effects of extreme cold on tumor tissues. Excessive cold causes intracellular and extracellular ice crystals to form in the affected tissue. These crystals damage intracellular organelles, especially mitochondria. The most lethal effect is the formation of intracellular ice crystals. This effect results from fast freezing and slow thawing cycles. In clinical practice, cryotherapy is used as an endobronchial treatment method capable of destroying tumor cells at a depth of 10 mm with a rigid probe and at a depth of 3 mm with a flexible probe.

The investigators investigated the treatment and long-term follow-up results of patients who underwent cryotherapy to the site of origin on the airway wall after the luminal part of the symptomatic endobronchial hamartomas was removed by interventional bronchoscopic methods. We aimed to determine the benefit of cryotherapy to conventional endobronchial debulking at the sites of origin of hamartomas.

Material and Methods:

General anesthesia was administered by an intravenous anesthesia technique. Patients were intubated with a rigid bronchoscope (Effer-Dumon, 11 mm diameter, 43 cm length, Efer Endoscopy, Marseille, France). Debulking procedures were performed by mechanical tumor resection (MTR) using the tip of the rigid bronchoscope, rigid pliers or argon plasma coagulation assisted MTR (ERBE ICC 200/APC 300 electrosurgical unit, rigid APC probe, 50 cm length, 2.3 mm diameter; ERBE, Medizintechnik, GmbH, Tübingen, Germany) or cryorecanalization (ERBOKRYO® CA unit, ERBE flexible cryoprobe 2.4 mm diameter, 90 cm length or ERBE rigid cryoprobe 3 mm diameter, 53 cm length; ERBE, Medizintechnik, GmbH, Tübingen, Germany) or electrocautery - snare probe (Erbotom ICC 200 electrosurgical unit ERBE, Medizintechnik GmbH, Tübingen, Germany and Electrosurgical snare probe SD-7C-1, loop diameter 23 mm, length 1050 mm, Olympus EndoTherapy, Tokyo, Japan). An innovation of study was that cryotherapy (Using the same equipment as cryorecanalization) was performed in the regions where the lesions originated after debulking.

Descriptive statistics were expressed as the mean ± standard deviation for intermittent and continuous numerical variables, and categorical variables were expressed as number of cases and "(%)".

This study has been approved by the local ethics committee. Informed consent was obtained from all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic endobronchial hamartomas treated by interventional bronchoscopic methods.

Exclusion Criteria:

* Patients with coagulation anomalies or low platelet counts, pregnancy, or who were younger than 18 years of age and those who did not sign the informed consent were excluded from the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Recurrences | 36 months
  Follow up recurrences

IPD SHARING:
Plan to Share IPD: No